CLINICAL TRIAL: NCT04509323
Title: A Randomized, Controlled, Single-center Clinical Study of Huperzine A in the Treatment of Brain Injury in Patients With Hypertensive Cerebral Hemorrhage
Brief Title: Clinical Study of Huperzine A in the Treatment of Patients With Hypertensive Cerebral Hemorrhage
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Jiangsu Famous Medical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: FM-P5-2020020501
Record Dates: First submitted 2020-07-22; First posted 2020-08-12 (Actual); Last update posted 2020-08-12 (Actual); Status verified 2020-08

CONDITIONS: Neurosensory Disorder
MeSH Terms: conditions — Sensation Disorders | interventions — huperzine A; Injections

STUDY DESIGN:
Intervention Model Description: Patients with hypertensive basal ganglia cerebral hemorrhage
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental：Huperzine A for Injection+Basic treatment (Experimental): Huperzine A for Injection: Dissolve each bottle with 2ml sterile water for injection and inject into muscle, the course of treatment is 14 days； Basic treatment：Control blood pressure; prevent continued bleeding; prevent and treat gastrointestinal bleeding; decide whether to perform dehydration treatment according to the condition to reduce cerebral edema; prevent infection, prevent various complications, etc.; routine rehabilitation training.
  Interventions: Drug: Huperzine A for Injection
- Control：Basic treatment (No Intervention): Basic treatment：Control blood pressure; prevent continued bleeding; prevent and treat gastrointestinal bleeding; decide whether to perform dehydration treatment according to the condition to reduce cerebral edema; prevent infection, prevent various complications, etc.; routine rehabilitation training.

INTERVENTIONS:
Drug: Huperzine A for Injection — Give the patient one intramuscular injection (0.2mg) of Huperzine A of injection once a day for 14 days
  Arms: Experimental：Huperzine A for Injection+Basic treatment

SUMMARY:
1. To evaluate the effectiveness of Huperzine A injection in the treatment of brain injury in patients with hypertensive cerebral hemorrhage；
2. To evaluate the safety of Huperzine A injection in the treatment of brain injury in patients with hypertensive cerebral hemorrhage。

DETAILED DESCRIPTION:
A randomized, controlled, single-center, exploratory clinical research method was used. In the treatment plan, the experimental group used basic treatment + Huperzine A, and the control group only used basic treatment, with a total of 20 cases. To evaluate the effectiveness and safety of Huperzine A injection in the treatment of brain injury in patients with hypertensive cerebral hemorrhage.

ELIGIBILITY:
Inclusion Criteria:

1. Aged from 18 to 75 years old(including 18 and 75 years old), males or females;
2. First onset, clinical diagnosis of hypertensive intracerebral hemorrhage, and CT confirmed that the amount of hemorrhage is between 15ml-50ml, the bleeding site is the basal ganglia, the bleeding has not penetrated into the lateral ventricle, and non-surgical patients；
3. Those with obvious neurological dysfunction after the onset, 5≤GCS≤15 or NIHSS≥6；
4. Admission within 72 hours after the onset of the disease, and no significant enlargement of the hematoma within 24 hours after admission (hematoma enlargement ≤ 5ml)；
5. The patient/family knows and signs the informed consent form voluntarily.

Exclusion Criteria:

1. Cerebral hemorrhage caused by cerebral aneurysm, brain tumor, brain trauma, cerebral parasitic disease, cerebrovascular malformation, abnormal blood vessel network at the base of the brain, cerebral arteritis, blood disease, metabolic disorder and other diseases confirmed by examination;
2. Patients with enlarged hematoma found within 24 hours after admission (the volume of enlarged hematoma> 5ml);
3. Patients with simple transient ischemic attack, lacunar infarction, subarachnoid hemorrhage and ischemic cerebral infarction;
4. Patients who use anticoagulant drugs for a long time;
5. Patients with platelet count <100,000, INR>1.4 at admission and abnormal blood coagulation function;
6. The measured value of homocysteine at admission is higher than 15μmol/L;
7. Patients who need surgical treatment (including ventricular drainage);
8. Patients with severe primary diseases such as cardiovascular, liver (ALT or AST>1.5 times the upper limit of normal), kidneys (BUN>1.5 times the upper limit of normal and Cr>upper limit of normal), endocrine system and hematopoietic system;
9. Those who are allergic to protein and test drugs;
10. People who are dependent on drugs or alcohol;
11. Intended pregnancy or women of childbearing age with positive pregnancy test and lactating women;
12. Participated in other clinical trials within the past 3 months;
13. Patients considered by the investigator to be inappropriate to participate in clinical trials.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2020-08-03 (Estimated); Primary Completion 2021-02-28 (Estimated); Study Completion 2021-05-28 (Estimated)

PRIMARY OUTCOMES:
Extension of Glasgow Outcome Scale(GOSE) Scores at 90 days of treatment | At the 90-day
  At the 90-day follow-up of patients, the extended Glasgow Outcome Scale (GOSE) was used to assess and judge the difference in consciousness after stroke between the two groups. The scores of minimum values is 1, the maximum values is 8, whether higher scores mean a better outcome.

SECONDARY OUTCOMES:
Extension of Glasgow Outcome Scale(GOSE) Scores at 30 days of treatment | At the 30-day
  At the 30-day follow-up of patients, the extended Glasgow Outcome Scale (GOSE) was used to assess and judge the difference in consciousness after stroke between the two groups. The scores of minimum values is 1, the maximum values is 8, whether higher scores mean a better outcome.
Scores of Modified Rankin Scale(mRS) at 14 days of treatment | At the 14-day
  At 14 days of treatment, the two groups of patients were scored with scores of Modified Rankin Scale(mRS). The mRS score of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 5, whether higher scores mean a worse outcome.
Scores of Modified Rankin Scale(mRS) at 30 days of treatment | At the 30-day
  At 30 days of treatment, the two groups of patients were scored with scores of Modified Rankin Scale(mRS). The mRS score of the two groups were compared whether there were statistical differences.The scores of minimum values is 0, the maximum values is 5, whether higher scores mean a worse outcome.
Scores of Modified Rankin Scale(mRS) at 90 days of treatment | At the 90-day
  At 90 days of treatment, the two groups of patients were scored with scores of Modified Rankin Scale(mRS). The mRS score of the two groups were compared whether there were statistical differences.The scores of minimum values is 0, the maximum values is 5, whether higher scores mean a worse outcome.
Scores of National Institute of Health stroke scale(NIHSS) at 14 days of treatment | At the 14-day
  At 14 days of treatment, the two groups of patients were scored with scores of National Institute of Health stroke scale(NIHSS). The NIHSS score of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 42, whether higher scores mean a worse outcome.
Scores of National Institute of Health stroke scale(NIHSS) at 30 days of treatment | At the 30-day
  At 30 days of treatment, the two groups of patients were scored with scores of National Institute of Health stroke scale(NIHSS). The NIHSS score of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 42, whether higher scores mean a worse outcome.
Scores of National Institute of Health stroke scale(NIHSS) at 90 days of treatment | At the 90-day
  At 90 days of treatment, the two groups of patients were scored with scores of National Institute of Health stroke scale(NIHSS). The NIHSS score of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 42, whether higher scores mean a worse outcome.
Scores of the Barthelindex of ADL at 14 days of treatment | At the 14-day
  At 14 days of treatment, the two groups of patients were scored with scores of Barthelindex of ADL. The Barthelindex of ADL scores of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 100, whether higher scores mean a better outcome.
Scores of the Barthelindex of ADL at 30 days of treatment | At the 30-day
  At 30 days of treatment, the two groups of patients were scored with scores of Barthelindex of ADL. The Barthelindex of ADL scores of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 100, whether higher scores mean a better outcome.
Scores of the Barthelindex of ADL at 90 days of treatment | At the 90-day
  At 90 days of treatment, the two groups of patients were scored with scores of Barthelindex of ADL. The Barthelindex of ADL scores of the two groups were compared whether there were statistical differences. The scores of minimum values is 0, the maximum values is 100, whether higher scores mean a better outcome.
Complication rate | At the 90-day
  After 90 days of treatment, compare whether the incidence of complications (including epilepsy, hydrocephalus, infarction, rebleeding, pneumonia, gastrointestinal hemorrhage) between the two groups is statistically different

CONTACTS AND LOCATIONS:
Locations (1):
- The Fifth Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: Undecided